CLINICAL TRIAL: NCT06499194
Title: Health Expenses and Outcomes of the DASH Diet in Egyptian Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ola Abu hashima abd elwahab, Mohamed Hassan Street from Salah Salem Street, Beni-Suef, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DASH diet and hypertension
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hypertension,Essential
Keywords: DASH diet; hypertension; health expense
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Intervention Model Description: an Open-label parallel design prospective controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Participants will taken a medical history review, anthropometric assessments, and waist circumference measurements. Tests included hemoglobin levels, kidney and liver function tests, fasting blood glucose, and lipid profiles. Baseline antihypertensive medications will be recorded in an Excel sheet and taken DASH diet .
  Interventions: Other: DASH diet
- control group (Placebo Comparator): Participants will taken a medical history review, anthropometric assessments, and waist circumference measurements. Tests included hemoglobin levels, kidney and liver function tests, fasting blood glucose, and lipid profiles. Baseline antihypertensive medications will be recorded in an Excel sheet and without taken DASH diet .
  Interventions: Other: DASH diet

INTERVENTIONS:
Other: DASH diet — The Dietary Approaches to Stop Hypertension (DASH) diets rich in fruits and vegetables and reduced in saturated fat can lower the risk for high blood pressure and assist with blood pressure control in hypertensive persons

SUMMARY:
DASH diet can reduce hypertension and decrease health expenses

DETAILED DESCRIPTION:
Hypertension is a prevalent cardiovascular risk factor associated with adverse outcomes and obesity. Egypt's prevalence is 26.3%, exceeding rates in the U.S. and sub-Saharan Africa. Lifestyle interventions like the DASH diet effectively manage hypertension, offering a cost-effective alternative to pharmacological treatments. This study aims to assess the effects of the DASH diet on blood pressure, BMI, waist circumference, and fasting blood glucose, as well as its cost-effectiveness compared to pharmacological treatments. This open-label prospective controlled clinical trial was conducted in Esna Health Administration, Luxor Governorate. The FMREC of Beni-Suef University approved the study, which included 364 hypertensive patients aged 30-60. Exclusions were patients with severe comorbidities or those who declined participation. Measurements included height, weight, BMI, blood pressure, and laboratory tests. The intervention group received a DASH diet education program. Outcomes measured were blood pressure, BMI, waist circumference, weight, and fasting blood glucose at baseline and post-intervention. Our study demonstrates the significant benefits of the DASH diet in managing blood pressure, weight, and fasting blood glucose levels in the Egyptian population. The DASH diet substantially reduced systolic and diastolic blood pressure, with a notable decrease in the number of antihypertensive medications needed. Additionally, participants on the DASH diet experienced significant weight loss and reduced BMI and waist circumference compared to the control group. The economic implications of the DASH diet are also promising, with a notable decrease in the total cost of therapy due to reduced medication costs.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with primary hypertension (all stages) in the family medicine units of Esna Health Administration, located in Luxor Governorate.
* Individuals between the ages of 30 and 60, of both male and female genders.

Exclusion Criteria:

* • Patients with cancer and either hepatic failure or renal impairment.

  * Patients diagnosed with diabetes, metabolic illness, or terminal organ failure.
  * A patient with severe or malignant hypertension.
  * Individuals who decline to partake in our research.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 364 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
blood pressure | 9 month
  patient on DASH diet showing decrease on blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abolfotouh MA, Soliman LA, Abolfotouh SM, Raafat M. Knowledge and Practice of PHC Physicians toward the Detection and Management of Hypertension and Other CVD Risk Factors in Egypt. Int J Hypertens. 2011;2011:983869. doi: 10.4061/2011/983869. Epub 2011 Aug 11. PMID 21860783
- [Background] Akhlaghi M. Dietary Approaches to Stop Hypertension (DASH): potential mechanisms of action against risk factors of the metabolic syndrome. Nutr Res Rev. 2020 Jun;33(1):1-18. doi: 10.1017/S0954422419000155. Epub 2019 Jul 30. PMID 31358075
- [Background] Al-Smair A, Saadeh O, Saadeh A, Al-Ali A. Renovascular Compression by the Diaphragmatic Crus: A Case Report. Cureus. 2022 Apr 10;14(4):e24004. doi: 10.7759/cureus.24004. eCollection 2022 Apr. PMID 35547452
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Ancker OV, Wehland M, Bauer J, Infanger M, Grimm D. The Adverse Effect of Hypertension in the Treatment of Thyroid Cancer with Multi-Kinase Inhibitors. Int J Mol Sci. 2017 Mar 14;18(3):625. doi: 10.3390/ijms18030625. PMID 28335429